CLINICAL TRIAL: NCT06324344
Title: Transcutaneous Electrical Nerve Stimulation for Lower Extremity in Patients With Neurogenic Pain - A Proof Concept Randomized Clinical Trial
Brief Title: Transcutaneous Electrical Nerve Stimulation (TENS) for Chemotherapy Induced Peripheral Neuropathy (CIPN)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI moved to another institution
Sponsor: Baylor College of Medicine (Other)
Collaborators: NeuroMetrix, Inc. (Industry)
Responsible Party: Principal Investigator, Bijan Najafi, PhD, Professor of Surgery, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H-50753-B
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Results first posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Pain; Neuropathy
Keywords: Transcutaneous Electrical Nerve Stimulation; Quell
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Participants who satisfy the inclusion and exclusion criteria and sign the informed consent form will be randomly assigned into two groups in a 1:1 ratio. One group will utilize high-dose TENS therapy (Intervention group, AG); the other group will utilize low-dose TENS devices (Placebo group, PG).
  Both groups will receive their respective devices at the initial visit (Baseline) and will be asked to return in 4 weeks and 8 weeks for follow-up assessment.
  Throughout this 8-week period the participants may receive follow-up phone calls assessing their compliance. All subjects will keep their active device after completion of the 8-week study.
Who Masked: Participant, Care Provider
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention Group (Active Comparator): The intervention group will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy on a daily basis with a high-dose TENS device for 8 weeks.
  The high-dose TENS device elicits 1 hour of TENS per session. Subjects are instructed to complete at least 3 sessions per day. To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side on a weekly basis.
  Interventions: Device: High-Dose TENS
- Placebo Group (Placebo Comparator): The placebo group will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy on a daily basis with a low-dose TENS device for 8 weeks.
  The low-dose TENS device is identical to the high-dose TENS device in all respects except that it delivers 6 minutes of TENS therapy per session (10% out of 60 minutes). Subjects are instructed to complete at least 3 sessions per day. To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side on a weekly basis.
  Interventions: Device: Low-Dose TENS

INTERVENTIONS:
Device: High-Dose TENS — high-dose TENS device delivers 1 hour of TENS therapy per session.
  Other Names: High Dose TENS; Active
  Arms: Intervention Group
Device: Low-Dose TENS — low-dose TENS device delivers 6 minutes of TENS therapy per session.
  Other Names: Placebo
  Arms: Placebo Group

SUMMARY:
The purpose of this pilot study is to examine the acceptability and proof of concept effectiveness of a wireless Transcutaneous Electrical Nerve Stimulation (TENS) technology to address Chemotherapy Induced Peripheral Neuropathy (CIPN). Participants, who satisfy the inclusion and exclusion criteria and sign the informed consent form will be randomly assigned with ratio of 1:1 into two groups. The patients and clinicians will be blinded for group allocation. One group will utilize TENS high-dose devices (Intervention group, IG); the other group will utilize low-dose TENS devices (Placebo group, PG). The baseline measurements will be performed, and the patients will take the programmed device home for a duration of 8 weeks. Then, the patients will come back after four weeks (4W) and after 8 weeks (8W) for outcome assessment. The primary outcome will be pain. Secondary outcomes include: nerve conduction and velocity, vibration perception threshold, quality of life. Exploratory outcomes include gait assessment (gait speed, stride length, double stance, and gait steadiness), and balance.

DETAILED DESCRIPTION:
Chemotherapy and other cancer treatments can cause damage to the peripheral nerves mainly reflected in severe pain in the upper and/or lower extremities. Additional to pain, cancer treatment may cause loss of balance which affects motor capacity and is a major cause of poor quality of life. There are only minimally effective treatments for CIPN despite over 20 years of research. Few recent studies have suggested that exercise intervention could be effective to restore numbness and motor capacity loss because of CIPN. Unfortunately, conventional rehabilitation programs however suffer from poor adherence and those programs for supervised settings have limitation of access for those who live in the remote areas (e.g., rural area), or could be too frail to travel after chemotherapy. This raised a significant disparity for delivering an effective therapy for those who are living in remote areas or those who are too frail to travel. Therefore, will test Quell® Transcutaneous Electrical Nerve Stimulation device developed by Neurometrix Inc. (Woburn, MA, USA), to mitigate the associated symptoms caused by CIPN. This device utilizes a wireless technology manageable through a smart phone application (Quell App) that also tracks symptom-status.

The investigators institution, Duncan Cancer Center (McNair Campus, Baylor College of Medicine St Luke's, Houston, Texas, USA) supervised by specialists in clinical and surgical oncology, has a high volume of patients that present with CIPN. Therefore, the investigators believe that this institution is a suitable place to perform this sub-study. The premise of this sub-study is that daily basis of TENS therapy could be effective to reduce pain, reduce numbness and improve both motor-capacity and mobility performance leading to improve quality of life in those who suffer from CIPN and have limited access to health care.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old willing and able to participate in study.
* Able to use an app via smart phone.
* Patients with Chemotherapy Induced Peripheral Neuropathy (CIPN) grades II and III.
* Have undergone chemotherapy with a drug known to cause neurotoxicity.
* Have finished chemotherapy ≥1 month, and still experiences CIPN.

Exclusion Criteria:

* Pregnancy or Lactation.
* Nerve Block a week prior to enrollment.
* Peripheral Sensory Neuropathy Grade I and IV.
* Patients applying ointments to the lower extremities.
* Patients with electrical implanted devices such as pacemakers.
* Patients with lower extremity wounds/history of minor/major amputation.
* Planning to undergo any type of chemotherapy in the next 3 months.
* Neuropathy derived from uncontrolled Diabetes Mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- High-Dose TENS: The intervention group will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy on a daily basis with a high-dose TENS device for 8 weeks.
  The high-dose TENS device elicits 1 hour of TENS per session. Subjects are instructed to complete at least 3 sessions per day. To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side on a weekly basis.
  High-Dose TENS: high-dose TENS device delivers 1 hour of TENS therapy per session.
- Low-Dose TENS: The Low-Dose TENS group will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy on a daily basis with a low-dose TENS device for 8 weeks.
  The low-dose TENS device is identical to the high-dose TENS device in all respects except that it delivers 6 minutes of TENS therapy per session (10% out of 60 minutes). Subjects are instructed to complete at least 3 sessions per day. To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side on a weekly basis.
  Low-Dose TENS: low-dose TENS device delivers 6 minutes of TENS therapy per session.
Period: Overall Study
Arm/Group | High-Dose TENS | Low-Dose TENS
Started | 5 | 5
Completed | 5 | 4
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: The intervention group will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy on a daily basis with a high-dose TENS device for 8 weeks.
  The high-dose TENS device elicits 1 hour of TENS per session. Subjects are instructed to complete at least 3 sessions per day. To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side on a weekly basis.
  High-Dose TENS: high-dose TENS device delivers 1 hour of TENS therapy per session.
- Placebo Group: The placebo group will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy on a daily basis with a low-dose TENS device for 8 weeks.
  The low-dose TENS device is identical to the high-dose TENS device in all respects except that it delivers 6 minutes of TENS therapy per session (10% out of 60 minutes). Subjects are instructed to complete at least 3 sessions per day. To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side on a weekly basis.
  Low-Dose TENS: low-dose TENS device delivers 6 minutes of TENS therapy per session.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Placebo Group | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11.70) | 64 (3.51) | 60 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27 (2.80) | 38 (7.26) | 32 (7.37)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Level at 8 Weeks From Baseline
Description: Pain was assessed using Item 9 of the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30, version 3), which ranges from 1 ("not at all" experiencing pain) to 4 ("very much" experiencing pain). The percentage change from baseline to week 8 was reported, with negative values indicating a reduction in pain and positive values indicating an increase in pain.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | High-Dose TENS | Low-Dose TENS
Number analyzed (Participants) | 5 | 4
Percent change | -18.33 (15.28) | 25 (0)

2. Secondary Outcome: Vibration Perception Threshold at 8 Weeks
Description: Change in Vibration Perception Threshold (VPT) will be assessed using the Neuro Touch device (Yostra Labs, Bengaluru, Karnataka, India). Measurements will be taken on the big toe of the participants' left and right feet to determine the minimum vibration intensity required to perceive sensation. VPT values range from 0 to 50 volts, with higher values indicating greater numbness.
Time Frame: week 8
Measure: Mean (Standard Deviation); unit: volts
Groups:
- High-Dose TENS: The intervention group (High-Dose TENS) will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy on a daily basis with a high-dose TENS device for 8 weeks.
  The high-dose TENS device elicits 1 hour of TENS per session. Subjects are instructed to complete at least 3 sessions per day. To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side on a weekly basis.
  High-Dose TENS: high-dose TENS device delivers 1 hour of TENS therapy per session.
- Low-Dose TENS: Low-Dose TENS group will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy on a daily basis with a low-dose TENS device for 8 weeks.
  The low-dose TENS device is identical to the high-dose TENS device in all respects except that it delivers 6 minutes of TENS therapy per session (10% out of 60 minutes). Subjects are instructed to complete at least 3 sessions per day. To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side on a weekly basis.
  Low-Dose TENS: low-dose TENS device delivers 6 minutes of TENS therapy per session.
Arm/Group | High-Dose TENS | Low-Dose TENS
Number analyzed (Participants) | 5 | 4
volts
  Right foot | 9.5 (5.4) | 16.2 (7.3)
  Left foot | 8.2 (9.5) | 17.2 (7.7)

3. Secondary Outcome: Quality of Life at 8 Weeks
Description: Quality of Life will be assessed using the European Organization for Research and Treatment in Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQC 30 ). It consists of 30 items divided into three main subscales: functional, symptom, and global health. Each subscale provides a comprehensive view of the patient's health and well-being.
  The Functional Scale measures physical, role, emotional, cognitive, and social functioning, with scores ranging from 0 to 100; higher scores indicate better functioning. The Symptom Scale evaluates cancer-related symptoms like fatigue, pain, and nausea, where higher scores (0-100) indicate greater symptom severity.
  The Global Health Scale assesses overall quality of life and general health, also scored from 0 to 100, with higher scores reflecting better health and well-being. These subscales provide critical insights for evaluating the impact of cancer and its treatment on patients.
Time Frame: week 8
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- High-dose TENS: The intervention group (High-dose TENS ) will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy on a daily basis with a high-dose TENS device for 8 weeks.
  The high-dose TENS device elicits 1 hour of TENS per session. Subjects are instructed to complete at least 3 sessions per day. To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side on a weekly basis.
  High-Dose TENS: high-dose TENS device delivers 1 hour of TENS therapy per session.
- Low-dose TENS: The placebo group (Low-dose TENS) will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy on a daily basis with a low-dose TENS device for 8 weeks.
  The low-dose TENS device is identical to the high-dose TENS device in all respects except that it delivers 6 minutes of TENS therapy per session (10% out of 60 minutes). Subjects are instructed to complete at least 3 sessions per day. To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side on a weekly basis.
  Low-Dose TENS: low-dose TENS device delivers 6 minutes of TENS therapy per session.
Arm/Group | High-dose TENS | Low-dose TENS
Number analyzed (Participants) | 5 | 4
score on a scale
  Functional scale | 72 (17.8) | 56 (24.3)
  Symptom scale | 61 (25.04) | 57 (21.9)
  Global Health | 33 (10.5) | 23 (7.2)

4. Other Pre Specified Outcome: Sural Nerve Conduction Velocity at 8 Weeks
Description: Sural nerve conduction velocity will be evaluated using the DPNCheck® device (Neurometrix, Woburn, MA, USA). The device is placed on the lateral portion of the patient's lower extremity and sends non-invasive electrical stimulation through the sural nerve to measure conduction velocity and amplitude. Conduction velocity is measured in meters per second (m/s), with normal values being greater than 40 m/s, while values below 40 m/s indicate slowed nerve signal transmission.
Time Frame: week 8
Population: Only 2 subjects out of five in the High-Dose TENS group and three subjects out of 4 in the Low-Dose TENS group completed this test.
Measure: Mean (Standard Deviation); unit: meters per second
Groups:
- High-Dose TENS: The High-Dose TENS group will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy on a daily basis with a high-dose TENS device for 8 weeks.
  The high-dose TENS device elicits 1 hour of TENS per session. Subjects are instructed to complete at least 3 sessions per day. To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side on a weekly basis.
  High-Dose TENS: high-dose TENS device delivers 1 hour of TENS therapy per session.
Arm/Group | High-Dose TENS | Low-Dose TENS
Number analyzed (Participants) | 2 | 3
meters per second | 48 (0) | 41.25 (13.1)

5. Other Pre Specified Outcome: Stride Time at 8 Weeks
Description: Stride time will be measured utilizing wearable sensors (LEGSys, Biosensics, MA) placed on both ankles, thighs and waist. The patient will be asked to walk for 30 feet in a normal pace. The unit is second and higher values indicate slower gait.
Time Frame: week 8
Population: Only 4 out of 5 participants in the High-Dose TENS group completed this test
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- High-dose TENS: The intervention group (high-dose TENS group) will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy on a daily basis with a high-dose TENS device for 8 weeks.
  The high-dose TENS device elicits 1 hour of TENS per session. Subjects are instructed to complete at least 3 sessions per day. To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side on a weekly basis.
  High-Dose TENS: high-dose TENS device delivers 1 hour of TENS therapy per session.
- Low-dose TENS: The placebo group (low-dose TENS group) will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy on a daily basis with a low-dose TENS device for 8 weeks.
  The low-dose TENS device is identical to the high-dose TENS device in all respects except that it delivers 6 minutes of TENS therapy per session (10% out of 60 minutes). Subjects are instructed to complete at least 3 sessions per day. To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side on a weekly basis.
  Low-Dose TENS: low-dose TENS device delivers 6 minutes of TENS therapy per session.
Arm/Group | High-dose TENS | Low-dose TENS
Number analyzed (Participants) | 4 | 4
seconds | 1.11 (.07) | 1.35 (.34)

6. Other Pre Specified Outcome: Cadence at 8 Weeks
Description: Cadence will be measured utilizing wearable sensors (LegSys, Biosensics, MA) placed on both ankles, thighs and waist. The patient will be asked to walk for 30 feet in a normal pace. The number is steps per minute, higher values indicate faster speed.
Time Frame: week 8
Measure: Mean (Standard Deviation); unit: steps/min
Groups:
- High-dose TENS: The intervention (high-dose TENS) group will be undergoing Transcutaneous Electrical Nerve Stimulation (TENS) therapy on a daily basis with a high-dose TENS device for 8 weeks.
  The high-dose TENS device elicits 1 hour of TENS per session. Subjects are instructed to complete at least 3 sessions per day. To deliver TENS, a band strap with hydrogel pads will be placed around the calf muscle of one lower-extremity alternating to the other side on a weekly basis.
  High-Dose TENS: high-dose TENS device delivers 1 hour of TENS therapy per session.
Arm/Group | High-dose TENS | Low-dose TENS
Number analyzed (Participants) | 4 | 4
steps/min | 108 (6.4) | 93 (19.0)

7. Other Pre Specified Outcome: Double-support Phase at 8 Weeks
Description: The double-support phase of gait will be measured utilizing wearable sensors (LEGSys, Biosensics, MA) placed on both ankles, thighs and waist. The patient will be asked to walk for 30 feet in a normal pace.
  The percentage of time the patient spends in the double support phase during the gait cycle will be recorded. Higher value indicates worst gait performance
Time Frame: week 8
Measure: Mean (Standard Deviation); unit: percentage of gait cycle
Arm/Group | High-dose TENS | Low-dose TENS
Number analyzed (Participants) | 4 | 4
percentage of gait cycle | 22.0 (2.3) | 29.1 (15.9)

8. Other Pre Specified Outcome: Balance at 8 Weeks
Description: Balance will be measured utilizing wearable sensors (BalaneSense, Biosensics, MA) placed on both ankles, thighs and waist. The patient will be asked to stand for 30 seconds with their eyes opened, then with their eyes closed. Center of Mass sway Area will be obtained from the hip and ankle motion. The unit is cm2 and higher value indicates poor balance. The center of mass sway was reported for eyes-closed condition.
Time Frame: week 8
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | High-dose TENS | Low-dose TENS
Number analyzed (Participants) | 4 | 4
cm2 | .84 (.244) | 2.36 (2.38)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Intervention Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT06324344/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT06324344/ICF_001.pdf